CLINICAL TRIAL: NCT06822348
Title: Short-term Effects of Osteopathic Manipulations on Heart Rate Variability in Lung Cancer Patients - A Randomized Pilot Study (OSTEOCAN2)
Brief Title: Short-term Effects of Osteopathic Manipulations on Heart Rate Variability in Lung Cancer Patients - A Randomized Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Duffaut - Avignon (Other)
Collaborators: Institut de Formation en Ostéopathie du Grand Avignon - IFO-GA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSTEOCAN2
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: osteopathy; heart rate variability; quality of life
MeSH Terms: conditions — Lung Neoplasms | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: 80 patients will be included, these patients will be randomized into two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Behavioral: Quality of life assessment; Behavioral: Anxiety assessment; Other: Heart rate variability assessment
- Osteopathy group (Experimental)
  Interventions: Other: Osteopathic treatment; Behavioral: Quality of life assessment; Behavioral: Anxiety assessment; Other: Heart rate variability assessment

INTERVENTIONS:
Other: Osteopathic treatment — Osteopathic manipulation
  Arms: Osteopathy group
Behavioral: Quality of life assessment — EORTC FA-12 questionnaire
Behavioral: Anxiety assessment — STAI-Y-A and STAI-Y-B questionnaire assessment
Other: Heart rate variability assessment — rMSSD (root mean square of successive R-R intervals), SDNN (standard deviation of all NN intervals), HF (high frequencies), LF (low frequencies), LF/HF ratio, Heart rate deceleration capacity, Heart rate acceleration capacity, Heart rate (bpm).

SUMMARY:
In France, the number of new cancer cases each year is rising steadily, while the number of deaths, although falling, is still around 157,000, including 23,000 from lung cancer alone. According to the French National Cancer Institute, there are three main methods of treating cancer: chemotherapy, radiotherapy and surgery. In recent years, new therapies have been developed, notably with the advent of immunotherapy and targeted therapies. On the other hand, although non-medical interventions (NMIs) such as osteopathy are recognized as improving the quality of life of cancer patients, there has been little research into their contribution when combined with conventional therapies.

Studies have shown a link between the vagus nerve and cancer. Through its actions, the vagus nerve regulates homeostasis and immunity at local and regional levels, reducing systemic inflammation but maintaining local inflammation, which has an anti-tumour effect. At the same time, vagus nerve stimulation increases heart rate variability, which, when increased, is associated with improved vital prognosis in cancer patients. This stimulation can be achieved using a number of common, non-invasive osteopathic techniques.

To date, no study has shown an objective and definitive link between vagus nerve stimulation and improved vital prognosis. However, several studies show that vagus nerve activity may be related to prognosis in cancer patients through regulation of HRV and possibly inflammation. Osteopathic manipulation to stimulate the vagus nerve could therefore have an effect on HRV. Improved HRV could therefore indirectly improve the prognosis of cancer patients. The first step is to test this clinical hypothesis: does osteopathic manipulation stimulate the vagus nerve in cancer patients? This will be done by measuring heart rate variability using rMSSD, the metric most representative of vagal tone.

This randomized single-center pilot study will investigate the short-term effect of vagus nerve stimulation using osteopathic techniques on heart rate variability in lung cancer patients. Our hypothesis is that stimulation of the vagus nerve by gentle, non-invasive osteopathic manipulation would increase vagal tone and therefore improve HRV and quality of life in the short term, but also reduce anxiety experienced at the time of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stage 4 lung cancer.
* WHO stage ≤ to 2.
* Dyspnea grade ≤ 2 on the mMRC scale (modified Medical Research Council)
* Patient undergoing chemotherapy for the first time
* Patient with less than 5% artifact rate during rMSSD measurement.
* Patient with SDNN less than 70 ms.
* Voluntary patient who has signed the informed consent form.
* No contraindications to osteopathic manipulation.

Exclusion Criteria:

* Patient with unilateral or bilateral vagotomy.
* Patient with cardiac arrhythmia.
* Patient undergoing treatment influencing cardiac rhythm (anti-arrhythmic drugs, beta-blockers, etc.)
* Patient with relapsed cancer already treated with chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of heart rate variability. | At baseline and before the first chemotherapy session
  rMSSD (root mean square of successive R-R intervals).

SECONDARY OUTCOMES:
Assessment of heart rate variability. | At baseline and before the first chemotherapy session
  SDNN (standard deviation of all NN intervals, measured in milliseconds).
Assessment of heart rate variability. | At baseline and before the first chemotherapy session
  HF (high frequencies, measured in milliseconds squared).
Assessment of heart rate variability. | At baseline and before the first chemotherapy session
  LF (low frequencies, measured in milliseconds squared).
Assessment of heart rate variability. | At baseline and before the first chemotherapy session
  LF/HF ratio (a low ratio could indicate parasympathetic dominance).
Assessment of heart rate variability. | At baseline and before the first chemotherapy session
  Heart rate deceleration capacity (measured in milliseconds).
Assessment of heart rate variability. | At baseline and before the first chemotherapy session
  Heart rate acceleration capacity (measured in milliseconds).
Assessment of heart rate variability. | At baseline and before the first chemotherapy session
  Heart rate (measured in beats per minute).
Osteopathic testing of somatic dysfunctions. | Before the first chemotherapy session
  Number of osteopathic vagus nerve dysfunctions.
Assessment of quality of life. | At baseline and before the second chemotherapy session
  EORTC QLQ-FA12 questionnaire (minimum = 0, maximum = 100, higher score means better outcome).
Anxiety assessment | At baseline
  State-Trait Anxiety Inventory : STAI-Y-B questionnaire (minimum = 20, maximum = 80, higher score means higher level of anxiety)
Anxiety assessment | Before the first chemotherapy session
  State-Trait Anxiety Inventory : STAI-Y-A questionnaire (minimum = 20, maximum = 80, higher score means higher level of anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Pierrick Martinez, Osteopath, Principal Investigator — Institut de Formation en Ostéopathie du Grand Avignon - IFO-GA
Locations (1):
- Centre Hospitalier d'Avignon, Hôpital Henri Duffaut, Avignon, France